CLINICAL TRIAL: NCT01600014
Title: Ingenol Mebutate Gel, 0.015% Repeat Use for Multiple Actinic Keratoses on Face and Scalp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0041-22; 2011-005018-13 (EudraCT Number)
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2016-04

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ingenol mebutate gel, 0.015% (Active Comparator): Topical field treatment once daily for 3 consecutive days on the face or scalp
  Interventions: Drug: Ingenol mebutate gel, 0.015%
- Vehicle gel (Placebo Comparator): Topical field treatment once daily for 3 consecutive days on the face or scalp
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: Ingenol mebutate gel, 0.015% — Topical field treatment once daily for 3 consecutive days within a 25 cm2 treatment area on the face or scalp of AKs present or emerging after an initial treatment with ingenol mebutate gel, 0.015%
  Arms: Ingenol mebutate gel, 0.015%
Drug: Vehicle gel — Topical field treatment once daily for 3 consecutive days within a 25 cm2 treatment area on the face or scalp of AKs present or emerging after an initial treatment with ingenol mebutate gel, 0.015%
  Arms: Vehicle gel

SUMMARY:
The purpose of the study is to demonstrate that ingenol mebutate gel is efficacious in treating Actinic Keratoses (AKs) present 8 weeks after initial field treatment or emerging in a previously cleared field.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide informed consent
* Subjects with 4 to 8 clinically typical, visible and discrete AKs within a contiguous 25 cm2 treatment area on the face or scalp
* Subject at least 18 years of age
* Female subjects must be of either:

  * Non-childbearing potential, i.e. post-menopausal or have a confirmed clinical history of sterility (e.g. the subject is without a uterus) or,
  * Childbearing potential, provided there is a confirmed negative urine pregnancy test prior to study treatment, to rule out pregnancy
* Female subjects of childbearing potential must be willing to consent to using highly effective methods of contraception

Exclusion Criteria:

* Location of the selected treatment area:

  * on any location other than the face or scalp
  * on the periorbital skin
  * within 5 cm of an incompletely healed wound
  * within 10 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC)
* Prior treatment with ingenol mebutate gel on face or scalp (previous treatment on trunk and extremities acceptable)
* Selected treatment area lesions that have atypical clinical appearance
* History or evidence of skin conditions other than the trial indication that would interfere with evaluation of the trial medication in the selected treatment area
* Anticipated need for hospitalization or out-patient surgery prior to Day 15 in the first treatment cycle
* Known sensitivity or allergy to any of the ingredients in ingenol mebutate gel
* Presence of sunburn within the selected treatment area
* Current enrollment or participation in a clinical trial within 30 days of entry into this study
* Subjects previously entered first treatment in the trial
* Female subjects who are breastfeeding
* Subjects who are institutionalised by court order or by the local authority
* In the opinion of the investigator, the subject is unlikely to comply with the Clinical Study Protocol

Prohibited Therapies and/or Medications within 2 weeks prior to Day 1

* Cosmetic or therapeutic procedures within 2 cm of the selected treatment area
* Use of keratolytic topical therapeutic products within 2 cm of the selected treatment area
* Use of topical medicated creams, ointments, lotions gels, foams or sprays within 2 cm of the selected treatment area; artificial tanners: within 5 cm of the selected treatment area

Prohibited Therapies and/or Medications: within 4 weeks prior to Day 1

* Treatment with immunomodulators, cytotoxic drugs or interferon /interferon inducers
* Treatment with systemic medications that suppress the immune system
* Treatment/therapy with ultraviolet light A (UVA) or ultraviolet light B (UVB)

Prohibited Therapies and/or Medications within 8 weeks prior to Day 1

* Treatment with 5-fluorouracil (5-FU), imiquimod, diclofenac sodium, or photodynamic therapy: within 2 cm of the selected treatment area

Prohibited Therapies and/or Medications within 6 months prior to Day 1

* Use of systemic retinoids or biologic/monoclonal antibody therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, MD, Principal Investigator — University Hospital Tuebingen
Locations (13):
- St John of God Dermatology, Subiaco, Australia
- Canada (9):
  - Stratica Medical, Edmonton, Alberta
  - Skin Care Centre, Vancouver, British Columbia
  - Dermadvances Research, Winnipeg, Manitoba
  - Durondel C.P. Inc./Dermatology Clinic, Moncton, New Brunswick
  - UltraNova Skincare, Barrie, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique, Québec, Quebec
- CHU de Nantes, Nantes, Loire-Atlantique 6, France
- Universitätsklinikum Tübingen, Tübingen, Germany
- Central Manchester University Hosptial, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 04-Jun-2012 Last Subject Last Visit: 05-Feb-2014
Pre-assignment Details: A total of 463 subjects were enrolled, 13 of whom were screening failures. 450 subjects were allocated to open label treatment with ingenol mebutate gel (1st cycle) and subsequently administered a 2nd cycle in a randomised vehicle controlled setting, if eligible for repeat use
Groups:
- Ingenol Mebutate Gel, 0.015% (1st & 2nd Cycle): Open label topical field treatment once daily for 3 consecutive days with ingenol mebutate 0.015% gel (1st cycle) within a 25 cm^2 treatment area on the face or scalp, followed by observation and/or repeat use (2nd cycle) once daily for 3 consecutive days with ingenol mebutate 0.015% gel of the same treatment area, in a randomised, controlled, double-blind setting, at Week 8 (field recalcitrant subgroup) or Week 26 or Week 44 (field recurrent subgroup) with follow-up until Week 52
- Vehicle Gel (2nd Cycle): Open label topical field treatment once daily for 3 consecutive days with mebutate 0.015% gel (1st cycle) within a 25 cm^2 treatment area on the face or scalp, followed by observation and/or repeat use (2nd cycle) once daily for 3 consecutive days with vehicle gel of the same treatment area, in a randomised, controlled, double-blind setting, at Week 8 (field recalcitrant subgroup) or Week 26 or Week 44 (field recurrent subgroup) with follow-up until Week 52
Period: 1. Cycle & Observation Period D1 to W52
Arm/Group | Ingenol Mebutate Gel, 0.015% (1st & 2nd Cycle) | Vehicle Gel (2nd Cycle)
Started | 450 (Subjects completing W52 without having been administered a 2nd cycle are counted as completers.) | 0
Completed | 162 | 0
Not Completed | 288 | 0
Not completed — Withdrawal by Subject | 24 | 0
Not completed — Included in 2nd cycle | 203 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Other | 27 | 0
Not completed — Exclusion Criteria Emerging during Study | 14 | 0
Not completed — Protocol Violation | 6 | 0
Not completed — Lost to Follow-up | 8 | 0
Period: 2. Cycle Recalcitrant Subgroup W8 to W52
Arm/Group | Ingenol Mebutate Gel, 0.015% (1st & 2nd Cycle) | Vehicle Gel (2nd Cycle)
Started | 92 | 49
Completed | 80 | 39
Not Completed | 12 | 10
Not completed — Death | 1 | 2
Not completed — Other | 1 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 5 | 0
Not completed — Exclusion Criteria Emerging during Study | 1 | 1
Not completed — Lost to Follow-up | 1 | 3
Period: 2. Cycl Recurrent Subgroup W26/44 to W52
Arm/Group | Ingenol Mebutate Gel, 0.015% (1st & 2nd Cycle) | Vehicle Gel (2nd Cycle)
Started | 42 | 20
Completed | 39 | 20
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ingenol Mebutate 0.015% Gel (1.& 2. Cycle): Open label topical field treatment once daily for 3 consecutive days with ingenol mebutate 0.015% gel (1st cycle) within a 25 cm^2 treatment area on the face or scalp, followed by observation and/or controlled repeat use (2nd cycle) treatment of recalcitrant or recurrent AK lesions
Arm/Group | Ingenol Mebutate 0.015% Gel (1.& 2. Cycle)
Number analyzed (Participants) | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 397

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Clearance of AKs 8 Weeks After Randomisation
Description: The complete clearance rates 8 weeks after randomisation was compared between ingenol mebutate gel, 0.015% and vehicle gel. Complete clearance was defined as no clinically visible AKs in the Selected Treatment Area (STA)
Time Frame: 8 weeks after randomisation
Measure: Number; unit: participants
Groups:
- Ingenol Mebutate Gel, 0.015% Field Recalcitrant Subgroup: Open label topical field treatment once daily for 3 consecutive days with ingenol mebutate 0.015% gel (1st cycle) within a 25 cm^2 treatment area on the face or scalp, followed by once daily for 3 consecutive days with ingenol mebutate 0.015% gel of the same treatment area (2nd cycle), in a randomised, controlled, double-blind setting, at Week 8 with follow-up until Week 52
- Vehicle Gel Field Recalcitrant Subgroup: Open label topical field treatment once daily for 3 consecutive days with mebutate 0.015% gel (1st cycle) within a 25 cm^2 treatment area on the face or scalp, followed by once daily for 3 consecutive days with vehicle gel of the same treatment area (2nd cycle), in a randomised, controlled, double-blind setting, at Week 8 with follow-up until Week 52
- Ingenol Mebutate Gel 0.015% Field Recurrent Subgroup: Open label topical field treatment once daily for 3 consecutive days with ingenol mebutate 0.015% gel (1st cycle) within a 25 cm^2 treatment area on the face or scalp, followed by once daily for 3 consecutive days with ingenol mebutate 0.015% gel of the same treatment area (2nd cycle), in a randomised, controlled, double-blind setting, at Week 26 or Week 44 with follow-up until Week 52
- Vehicle Gel Field Recurrent Subgroup: Open label topical field treatment once daily for 3 consecutive days with mebutate 0.015% gel (1st cycle) within a 25 cm^2 treatment area on the face or scalp, followed by once daily for 3 consecutive days with vehicle gel of the same treatment area (2nd cycle), in a randomised, controlled, double-blind setting, at Week 26 or Week 44 with follow-up until Week 52
Arm/Group | Ingenol Mebutate Gel, 0.015% Field Recalcitrant Subgroup | Vehicle Gel Field Recalcitrant Subgroup | Ingenol Mebutate Gel 0.015% Field Recurrent Subgroup | Vehicle Gel Field Recurrent Subgroup
Number analyzed (Participants) | 92 | 49 | 42 | 20
participants | 43 | 9 | 25 | 5
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel, 0.015% Field Recalcitrant Subgroup vs Vehicle Gel Field Recalcitrant Subgroup; The analysis type was superiority between groups. In total 141 subjects were included; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — Chi-square test for stratified data with a significance level of 5%. No adjustment for multiple tests was needed, due to the analyses were based on distinct subject groups; Cochran-Mantel-Haenszel ratio of clearance rates (Ingenol mebutate relative to Vehicle) adjusted for anatomical location and country; Risk Ratio (RR) = 2.44, 95% CI 2-sided [1.32 to 4.51]
Statistical Analysis 2: Comparison: Ingenol Mebutate Gel 0.015% Field Recurrent Subgroup vs Vehicle Gel Field Recurrent Subgroup; The analysis type was superiority between groups. In total 62 subjects were included; Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel ratio of clearance rates (Ingenol mebutate relative to Vehicle) adjusted for anatomical location and week of randomisation; Risk Ratio (RR) = 2.37, 95% CI 2-sided [1.07 to 5.25]

2. Secondary Outcome: Number of Participants With Complete Clearance Through to Month 12, Defined as no Clinically Visible AKs and no Lesions Treated in the Selected Treatment Area at Any Time From Last Treatment Cycle Through to Month 12
Description: The analysis was done separately for the field recalcitrant subgroup, the field recurrent subgroup, and overall for all treated subject (Analysis 1, 2, and 3, respectively)
Time Frame: From last treatment cycle through to Month 12
Measure: Number; unit: participants
Groups:
- Open Label Only (1st Cycle): Subjects only treated during 1st cycle (450 participants excluding 203 participants also included in the 2nd cycle)
- Ingenol Mebutate Gel, 0.015% Field Recalcitrant Subgroup; Vehicle Gel Field Recalcitrant Subgroup; Ingenol Mebutate Gel 0.015% Field Recurrent Subgroup; Vehicle Gel Field Recurrent Subgroup: See primary endpoint for previously defined description
Arm/Group | Open Label Only (1st Cycle) | Ingenol Mebutate Gel, 0.015% Field Recalcitrant Subgroup | Vehicle Gel Field Recalcitrant Subgroup | Ingenol Mebutate Gel 0.015% Field Recurrent Subgroup | Vehicle Gel Field Recurrent Subgroup
Number analyzed (Participants) | 247 | 92 | 49 | 42 | 20
participants | 124 | 17 | 2 | 13 | 3
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel, 0.015% Field Recalcitrant Subgroup vs Vehicle Gel Field Recalcitrant Subgroup; The analysis type was superiority between groups. In total 141 subjects were included; Test type: Superiority or Other; p = 0.016, Cochran-Mantel-Haenszel — A closed test procedure was chosen where the evaluation process stopped when the first non-significant results were observed thus securing that the overall significance level did not exceed 5% for multiple testing; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 4.41, 95% CI 2-sided [1.10 to 17.62]
Statistical Analysis 2: Comparison: Ingenol Mebutate Gel 0.015% Field Recurrent Subgroup vs Vehicle Gel Field Recurrent Subgroup; The analysis type was superiority between groups. In total 62 subjects were included; Test type: Superiority or Other; p = 0.10, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 2.24, 95% CI 2-sided [0.78 to 6.47]
Statistical Analysis 3: Comparison: Open Label Only (1st Cycle) vs Ingenol Mebutate Gel, 0.015% Field Recalcitrant Subgroup vs Ingenol Mebutate Gel 0.015% Field Recurrent Subgroup; Subjects randomised to vehicle were not included in the estimate of the overall clearance rate for the repeat-use regimen, from last treatment throught to Month 12. Instead, the subjects randomised to ingenol mebutate were given higher weights to reflect the hypothetical scenario where all randomised subjects were given active treatment during the repeat use cycle; Test type: Superiority or Other; Percent cleared subjects = 50.0, 95% CI 2-sided [44.0 to 56.1] — Estimation based on completers only

3. Secondary Outcome: The Change in AK Count From Randomisation to 8 Weeks After Randomisation
Description: The change in AK count from randomisation to 8 weeks after randomisation was determined for the field recalcitrant and the field recurrent subgroups
Time Frame: 8 weeks after randomisation
Measure: Mean (Standard Deviation); unit: AK count
Arm/Group | Ingenol Mebutate Gel, 0.015% Field Recalcitrant Subgroup | Vehicle Gel Field Recalcitrant Subgroup | Ingenol Mebutate Gel 0.015% Field Recurrent Subgroup | Vehicle Gel Field Recurrent Subgroup
Number analyzed (Participants) | 92 | 49 | 42 | 20
AK count | -1.41 (1.49) | -0.51 (1.65) | -1.52 (1.49) | -0.85 (0.99)
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel, 0.015% Field Recalcitrant Subgroup vs Vehicle Gel Field Recalcitrant Subgroup; The analysis type was superiority between groups. In total 141 subjects were included; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Analysed using ANCOVA adjusted for anatomical location, country and AK count at randomisation; Mean Difference (Net) = -0.88, 95% CI 2-sided [-1.38 to -0.38] — Using baseline observation carried forward (BOCF) as the imputation method
Statistical Analysis 2: Comparison: Ingenol Mebutate Gel, 0.015% Field Recalcitrant Subgroup vs Vehicle Gel Field Recalcitrant Subgroup; The analysis type was superiority between groups. In total 141 subjects were included; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Sensitivity analysis using complete cases; Mean Difference (Net) = -1.01, 95% CI 2-sided [-1.52 to -0.51] — Sensitivity analysis using complete cases
Statistical Analysis 3: Comparison: Ingenol Mebutate Gel 0.015% Field Recurrent Subgroup vs Vehicle Gel Field Recurrent Subgroup; The analysis type was superiority between groups. In total 62 subjects were included; Test type: Superiority or Other; p = 0.008, ANCOVA — Formal statistical significance could not be established because of the closed test procedure where the first secondary endpoint tested (12 months clearance) did not reach statistical significance in the recurrent subgroup; Analysed using ANCOVA adjusted for anatomical location, country and AK count at randomisation; Mean Difference (Net) = -0.69, 95% CI 2-sided [-1.19 to -0.19] — Using BOCF as the imputation method, the difference in the adjusted mean AK count between the ingenol mebutate and vehicle groups

ADVERSE EVENTS:
Time Frame: 8-week treatment periods (1st or 2nd cycle)
Groups:
- Ingenol Mebutate 0.015% Gel (1. Cycle): Open label topical field treatment once daily for 3 consecutive days with ingenol mebutate 0.015% gel within a 25 cm2 treatment area on the face or scalp
- Ingenol Mebutate 0.015% Gel (2. Cycle): Repeat use once daily for 3 consecutive days with ingenol mebutate 0.015% gel of the same treatment area (25 cm2 treatment area on the face or scalp) in a randomised, controlled, double-blind setting, at Week 8 (field recalcitrant subgroup) or Week 26 or Week 44 (field recurrent subgroup)
- Vehicle Gel (2. Cycle): Repeat use once daily for 3 consecutive days with vehicle gel of the same treatment area (25 cm2 treatment area on the face or scalp) in a randomised, controlled, double-blind setting, at Week 8 (field recalcitrant subgroup) or Week 26 or Week 44 (field recurrent subgroup)
Arm/Group | Ingenol Mebutate 0.015% Gel (1. Cycle) | Ingenol Mebutate 0.015% Gel (2. Cycle) | Vehicle Gel (2. Cycle)
Serious Adverse Events (participants affected / at risk) | 7/450 | 1/134 | 3/69
Other Adverse Events (participants affected / at risk) | 197/450 | 61/134 | 19/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ingenol Mebutate 0.015% Gel (1. Cycle) (N=450) | Ingenol Mebutate 0.015% Gel (2. Cycle) (N=134) | Vehicle Gel (2. Cycle) (N=69)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ingenol Mebutate 0.015% Gel (1. Cycle) (N=450) | Ingenol Mebutate 0.015% Gel (2. Cycle) (N=134) | Vehicle Gel (2. Cycle) (N=69)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (23) | 5 (11) | 6 (8)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (6) | 4 (6)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 21 (24) | 0 (0) | 2 (2)
Eyelid oedema (Eye disorders) | 17 (18) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 15 (16) | 0 (0) | 0 (0)
Application site pain (General disorders) | 62 (71) | 15 (19) | 0 (0)
Application site pruritus (General disorders) | 20 (20) | 7 (7) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 43 (51) | 21 (38) | 3 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.